CLINICAL TRIAL: NCT01580020
Title: An Open-label, Multi-center, 6-month Extension Study Comparing the Long-term Efficacy and Safety of Lucentis (Ranibizumab) Intravitreal Injections Versus Ozurdex (Dexamethasone) Intravitreal Implant in Patients With Visual Impairment Due to Macular Edema Following Branch Retinal Vein Occlusion (BRVO) or Central Retinal Vein Occlusion (CRVO) Who Have Completed the Respective Core Study (CRFB002EDE17 or CRFB002EDE18)
Brief Title: Extension Study to Compare Long-term Efficacy and Safety of Ranibizumab Intravitreal Injections Versus Dexamethasone Intravitreal Implant in Patients With RVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002EDE20; 2011-005045-13 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Retinal Vein Occlusion
Keywords: Macular Degeneration; Macular Edema; Retinal Vein Occlusion; Choroidal Neovascularization; Signs and Symptoms; Retinal Degeneration; Retinal Diseases; Eye Diseases; Venous Thrombosis Sensation Disorders; Dexamethasone acetate; Dexamethasone; Dexamethasone 21-phosphate; BB 1101; Anti-Inflammatory Agents; Therapeutic Uses; Vision, Low; Signs; Vision Disorders
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Degeneration; Macular Edema; Choroidal Neovascularization; Signs and Symptoms; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision, Low; Vision Disorders | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Arm A) (Experimental): The PRN injection scheme applied in the core study will also be followed during this extension study:
  Patients should be monitored monthly (starting at V1E) for VA and treatment is to be resumed when monitoring indicates loss of VA due to disease activity. Monthly injections should then be administered until stable VA is reached again for 3 consecutive monthly assessments (implying a minimum of 2 injections during stable VA). The interval between 2 doses should not be shorter than 1 month
  Interventions: Biological: RFB002
- Dexamethasone (Arm B) (Sham Comparator): A PRN re-treatment scheme will be applied for the Ozurdex arm during this extension study, i.e. patients may receive an implant at V1E or later as needed: Patients should be monitored monthly and if there is a decline from stable VA stability due to macular edema patients will receive another intravitreal implant. (700 µg; long acting release (LAR)) given that in the opinion of the investigator the patient would benefit from the re-treatment. However, a minimum period of 5 months in between implantations is required.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Biological: RFB002 — 0.5 mg/0.05 mL solution to be injected intravitreally. Ranibizumab was formulated as a sterile solution aseptically filled in a sterile glass vial. Each vial contained ranibizumab in an aqueous solution (pH 5.5) with histidine, trehalose and polysorbate 20.
  Arms: Ranibizumab (Arm A)
Drug: Dexamethasone — Ozurdex (Dexamethasone): intravitreal implant as per commercial label (700 µg Dexamethasone; Dexamethasone was formulated as a rod shaped implant to be inserted into the eye by an applicator. The implant as well as the respective applicator were suitable for single use only. Dexamethasone had to be stored according to label instructions and it had to be kept in a secure locked facility
  Arms: Dexamethasone (Arm B)

SUMMARY:
The study is intended to characterize the clinical benefit regarding safety and efficacy of a long term treatment with Lucentis in comparison with Ozurdex over an additional 6 months and a 3-month follow-up period, following the initial 6-month treatment in the respective core studies CRFB002EDE17 (NCT01396057) and CRFB002EDE18 (NCT01396083).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the core study assessments at month 6 of study CRFB002EDE17 or CRFB002EDE18, respectively

Exclusion Criteria:

* Patients who experienced an uncontrollable rise in IOP during the core study CRFB002EDE17 respectively CRFB002EDE18, i.e. IOP could not be decreased to a stable level of < 25mmHg.
* Use of other investigational drugs
* Current use or likely need of systemic medications known to be toxic to the lens, retina or optic nerve
* History of hypersensitivity to Ranibizumab or Ozurdex or any component of the ranibizumab respectively Ozurdey formulation
* Any type of advanced, severe or unstable disease or its treatment, that could interfere with evaluations or put the patient at special risk
* Women
* who were pregnant or breast feeding (pregnancy defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/mL)
* who were menstruating and capable of becoming pregnant* and not practicing a medically approved method of contraception (Pearl Index <1**)*** during and up to at least 4 weeks after the end of treatment. A negative pregnancy test (serum) for all women and for girls entering menarche was required with sufficient lead time before randomization

  * definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy

    * examples of particularly reliable methods with Pearl Index (PI) <1, according to guidelines of "Deutsche Gesellschaft für Gynäkologie und Geburtshilfe":

      * Combination pill with estrogen and gestagen (no mini-pill, PI=0.1-0.9)
      * Vaginal ring (NuvaRing®, PI=0.65 uncorr.; 0.4 corr.)
      * Contraceptive patch (EVRA®, PI= 0.72 uncorr.; 0.9 corr.)
      * Estrogen-free ovulation inhibitors (Cerazette®, PI=0.14)
      * Progestin-containing contraceptives (Implanon®, PI=0-0.08)
      * Injectable 3-month depot progestins (PI=0.3-1.4; 0.88 corr.)
      * Intra-uterine progestin device (Mirena®, PI=0.16)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- Germany (32):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Regensburg, Germany
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Rothenfelde
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg I. Br
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ingolstadt
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Sulzbach
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 140 patients with (BRVO) completed the core study CRFB002EDE17, and 127 patients with (CRVO) completed the core study CRFB002EDE18. 92 patients with BRVO and 83 patients with CRVO were enrolled into the extension study. A total of 175 patients (113 in the ranibizumab group and 62 in the dexamethasone group) were enrolled
Pre-assignment Details: The Full Analysis Sets (FAS) consisted of all patients from the FAS of the respective core study who had received at least one application of study treatment and had at least one post- baseline assessment for BCVA during the extension study. LOCF=last observation carried forward
Groups:
- Ranibizumab (BRVO): Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally
- Dexamethasone (BRVO); Dexamethasone (CRVO): A PRN re-treatment scheme will be applied for the Dexamethasone arm during this extension study, i.e. patients may receive an implant at V1E or later as needed. Intravitreal implant as per commercial label (700 μg Dexamethasone; long acting release (LAR) Minimum period of 5 months in between implantations was required.
- Ranibizumab (CRVO): Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitrally
Period: Overall Study
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Started | 52 | 40 | 61 | 22
Completed | 51 | 33 | 57 | 20
Not Completed | 1 | 7 | 4 | 2
Not completed — Lack of Efficacy | 0 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Administrative Problems | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab: Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally
- Dexamethasone: A PRN re-treatment scheme will be applied for the Dexamethasone arm during this extension study, i.e. patients may receive an implant at V1E or later as needed. Intravitreal implant as per commercial label (700 μg Dexamethasone; long acting release (LAR) Minimum period of 5 months in between implantations was required.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Dexamethasone | Total
Number analyzed (Participants) | 113 | 62 | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (9.9) | 63.3 (10.3) | 64.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 26 | 90
  Male | 49 | 36 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The number of participants who experienced Adverse events, serious AE and death
Time Frame: 6 months
Population: The Safety Set consisted of all patients from the safety sets of the respective core study who had received at least one application of study treatment and had at least one safety assessment during the extension study. Patients were analyzed according to treatment received.
Measure: Number; unit: Participants
Groups:
- Ranibizumab (CRVO): Injections consisted of 0.5 mg/0.05 ml solution to be injected intravitreally
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 61 | 22
Participants
  Adverse event | 35 | 28 | 45 | 16
  Serious adverse event | 2 | 3 | 6 | 1
  Death | 0 | 0 | 0 | 0

2. Secondary Outcome: Raw Mean Best Corrected Visual Acuity (BCVA) by Treatment Group
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. The range of BCVA (EDTRS) is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement
Time Frame: Baseline, 6 months and 12 months
Population: FAS consisted of all patients from the FAS of the respective core study who had received at least one application of study treatment and had at least one post- baseline assessment for BCVA during the extension study. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned.
Measure: Mean (Standard Deviation); unit: Letters read correctly
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 60 | 22
Letters read correctly
  Baseline | 56.8 (10.0) | 58.3 (10.8) | 53.8 (15.7) | 53.2 (16.1)
  Month 6 | 77.9 (10.6) | 69.2 (11.9) | 72.6 (13.5) | 64.1 (24.0)
  Month 12 | 79.0 (10.1) | 70.6 (13.9) | 72.6 (15.8) | 66.6 (22.3)

3. Secondary Outcome: Percentage of Patients Gaining / Losing ≥ 15 / 10 / 5 Letters at Month 12 Compared to Baseline
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who were gaining/losing ≥15, 10 or 5 more letters of visual acuity at month 12 as compared with baseline
Time Frame: 12 month
Population: Full Analysis Sets (FAS) consisted of all patients from the FAS of the respective core study who had received at least one application of study treatment and had at least one post- baseline assessment for BCVA during the extension study. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 60 | 22
Percentage of participants
  Gain≥15 letters | 80.8 | 50.0 | 58.3 | 45.5
  Gain ≥10 letters | 88.5 | 65.0 | 75.0 | 68.2
  Gain ≥5 letters | 100.0 | 80.0 | 86.7 | 77.3
  Loss of ≥15 letters | 0.0 | 7.5 | 0.0 | 4.5
  Loss of ≥10 letters | 0.0 | 10.0 | 0.0 | 4.5
  Loss of ≥5 letters | 0.0 | 10.0 | 3.3 | 4.5

4. Secondary Outcome: Change in Central Subfield Thickness (CSRT) From Baseline to Month 12
Description: High Resolution OCT was performed at every study visit by Spectral Domain OCT (if not available Time Domain OCT was acceptable) and the images were transferred to a digital video disc. These assessments were performed by trained and adequately qualified experts at the sites and prior to any study drug administration. CSFT is the average retinal thickness of the circular area with 1 mm diameter around the foveal center.
Time Frame: Baseline , Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 59 | 22
um | -288.1 (180.6) | -211.5 (199.3) | -374.6 (239.8) | -360.3 (260.2)

5. Secondary Outcome: Change of Foveal Center Point Thickness (FCPT) From Baseline to Month 12
Description: FCPT (foveal center point thickness) was assessed by central reading center to ensure error- corrected measurements of retinal thickness and volumes,
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 51 | 39 | 58 | 21
um | -341.8 (226.2) | -252.6 (197.9) | -439.4 (279.8) | -432.3 (245.8)

6. Secondary Outcome: Change in Mean Visual Function Questionnaire (VFQ-25)
Description: The VFQ-25 composite and subscale scores range from 0 to 100, a higher score indicating better functioning. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated improvement in quality of life due to vision function.
Time Frame: Baseline, 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 60 | 22
Scores on a scale
  Overall Composite | 8.1 (10.6) | 5.5 (11.3) | 9.1 (15.5) | 10.0 (15.9)
  General Health | -1.4 (15.2) | 6.3 (18.6) | 1.7 (18.9) | 5.7 (20.3)
  General Vision | 15.0 (16.7) | 9.5 (16.3) | 20.0 (17.7) | 13.6 (23.4)
  Ocular Pain | 5.3 (15.7) | 5.3 (13.8) | 4.2 (20.8) | 3.4 (15.0)
  Near Activities | 13.3 (18.9) | 10.8 (20.6) | 12.3 (20.5) | 12.3 (23.2)
  Distance Activities | 8.9 (17.5) | 5.6 (15.3) | 7.8 (18.3) | 8.3 (23.4)
  Social Functioning | 3.4 (16.8) | 2.2 (12.0) | 3.3 (16.7) | 2.8 (21.1)
  Mental Health | 10.2 (14.9) | 2.9 (20.4) | 10.7 (21.7) | 15.1 (18.3)
  Role Difficulties | 4.8 (26.8) | 10.6 (20.5) | 14.6 (29.9) | 24.4 (27.8)
  Dependency | 3.2 (9.2) | 0.4 (16.6) | 5.1 (16.7) | 4.4 (12.8)
  Driving (BRVO n=44,31) (CRVO n=42,16) | 11.7 (23.9) | 4.8 (21.3) | 14.2 (24.6) | 17.7 (25.1)
  Color Vision(BRVO n=52,39) | 0.5 (10.5) | 1.9 (10.6) | 0.4 (17.5) | -1.1 (14.4)
  Peripheral Vision(BRVO n=51,40) | 10.3 (24.1) | 6.9 (23.3) | 11.7 (25.0) | 14.8 (22.7)

7. Secondary Outcome: Change in SF-36 Summary Scores
Description: The SF-36 measures the impact of disease on overall quality of life and consists of eight subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score. Scores for each subscale range from 0 to 10, and the composite scores range from 0 to 100, with higher scores indicating better health. A positive change from Baseline score indicates improvement in quality of life.
Time Frame: Baseline, month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 60 | 22
Score on a scale
  Physical Component(BRVO n=50,39) (CRVO n=58,20) | 1.6 (5.0) | 0.2 (7.0) | -1.1 (8.2) | 1.3 (7.2)
  Mental Component (BRVO n=50,39) (CRVO n=58,20) | 3.3 (9.7) | 2.1 (13.2) | 2.1 (9.3) | 2.4 (12.4)

8. Secondary Outcome: Change in Euro Quality of Life Questionnaire (EQ-5D) VAS Summary Scores
Description: The Euro Quality of Life Questionnaire (EQ-5D) standardized instrument was utilized to measure health outcomes related to mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Participants self-rate their health on a visual, vertical analogue scale from 0 to 100 where the endpoints are labeled "Best imaginable health state" (100) and "worst imaginable health state" (0).
Time Frame: Baseline, month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 58 | 21
Score on a scale | 3.3 (15.2) | 2.6 (16.9) | 1.5 (16.4) | 0.2 (20.4)

9. Secondary Outcome: Time to the First Retreatment of Both Treatment Arms
Description: Time to the first retreatment
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Number analyzed (Participants) | 52 | 40 | 61 | 22
Days | 37 [3 to 56] | NA [328 to NA] — Not calculable because <50% of patients received re-treatment | 62 [5 to 67] | NA [309 to NA] — Not calculable because <50% of patients received re-treatment

ADVERSE EVENTS:
Description: The Safety Set consisted of all patients from the safety sets of the respective core study who had received at least one application of study treatment and had at least one safety assessment during the extension study. Patients were analyzed according to treatment received.
Arm/Group | Ranibizumab (BRVO) | Dexamethasone (BRVO) | Ranibizumab (CRVO) | Dexamethasone (CRVO)
Serious Adverse Events (participants affected / at risk) | 2/52 | 3/40 | 6/61 | 1/22
Other Adverse Events (participants affected / at risk) | 35/52 | 28/40 | 45/61 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (BRVO) (N=52) | Dexamethasone (BRVO) (N=40) | Ranibizumab (CRVO) (N=61) | Dexamethasone (CRVO) (N=22)
GLAUCOMA (Fellow eye) (Eye disorders) | 0 | 0 | 1 | 0
GLAUCOMA (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
IRIS NEOVASCULARISATION (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
MACULAR OEDEMA (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
OCULAR ISCHAEMIC SYNDROME (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
RETINAL DETACHMENT (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
VITREOUS HAEMORRHAGE (Study eye) (Eye disorders) | 0 | 0 | 1 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
SUBSTANCE ABUSE (Psychiatric disorders) | 0 | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (BRVO) (N=52) | Dexamethasone (BRVO) (N=40) | Ranibizumab (CRVO) (N=61) | Dexamethasone (CRVO) (N=22)
FACTOR V LEIDEN MUTATION (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
CATARACT (Study eye) (Eye disorders) | 0 | 3 | 2 | 1
CONJUNCTIVAL HAEMORRHAGE (Study eye) (Eye disorders) | 2 | 7 | 3 | 3
CONJUNCTIVAL HYPERAEMIA (Study eye) (Eye disorders) | 0 | 0 | 1 | 1
CONJUNCTIVAL IRRITATION (Study eye) (Eye disorders) | 1 | 2 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Study eye) (Eye disorders) | 0 | 1 | 0 | 1
DRY EYE (Fellow eye) (Eye disorders) | 2 | 1 | 0 | 0
DRY EYE (Study eye) (Eye disorders) | 3 | 1 | 0 | 0
EYE PAIN (Study eye) (Eye disorders) | 4 | 0 | 7 | 4
FOREIGN BODY SENSATION IN EYES (Study eye) (Eye disorders) | 0 | 1 | 4 | 0
GLAUCOMA (Study eye) (Eye disorders) | 0 | 1 | 1 | 1
LACRIMATION INCREASED (Study eye) (Eye disorders) | 6 | 2 | 2 | 2
MACULAR FIBROSIS (Study eye) (Eye disorders) | 0 | 0 | 2 | 0
MACULAR OEDEMA (Study eye) (Eye disorders) | 9 | 3 | 14 | 3
OCULAR DISCOMFORT (Study eye) (Eye disorders) | 2 | 4 | 1 | 0
OCULAR HYPERAEMIA (Study eye) (Eye disorders) | 7 | 3 | 4 | 3
PHOTOPSIA (Study eye) (Eye disorders) | 0 | 0 | 2 | 0
RETINAL EXUDATES (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
RETINAL ISCHAEMIA (Study eye) (Eye disorders) | 5 | 4 | 2 | 0
RETINAL OEDEMA (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
VISION BLURRED (Study eye) (Eye disorders) | 1 | 0 | 4 | 1
VISUAL ACUITY REDUCED (Study eye) (Eye disorders) | 4 | 4 | 8 | 1
VISUAL IMPAIRMENT (Study eye) (Eye disorders) | 0 | 0 | 1 | 1
VITREOUS DETACHMENT (Fellow eye) (Eye disorders) | 0 | 2 | 1 | 0
VITREOUS DETACHMENT (Study eye) (Eye disorders) | 2 | 2 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 2 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 2 | 2 | 0
CONJUNCTIVITIS (Study eye) (Infections and infestations) | 0 | 1 | 2 | 0
CYSTITIS (Infections and infestations) | 2 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 2 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 1 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 9 | 3 | 12 | 3
PERIODONTITIS (Infections and infestations) | 1 | 0 | 1 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 2 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
POST PROCEDURAL SWELLING (Study eye) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1
INTRAOCULAR PRESSURE DECREASED (Study eye) (Investigations) | 0 | 0 | 0 | 1
INTRAOCULAR PRESSURE INCREASED (Study eye) (Investigations) | 3 | 10 | 3 | 4
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 0 | 2 | 1 | 1
SCIATICA (Nervous system disorders) | 1 | 0 | 2 | 0
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety